CLINICAL TRIAL: NCT03674671
Title: Investigations on the Efficacy of Ketamine in Depression in Comparison to Electroconvulsive Therapy
Brief Title: Ketamine Versus Electroconvulsive Therapy in Depression
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient funding
Sponsor: University of Ottawa (Other)
Collaborators: McGill University (Other); Queen's University (Other); University Health Network, Toronto (Other); Ontario Shores Centre for Mental Health Sciences (Other)
Responsible Party: Principal Investigator, Pierre Blier, Endowed Chair and Director, Mood Disorders Research Unit, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REB2018007
Record Dates: First submitted 2018-07-06; First posted 2018-09-17 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Depressive Disorder, Major; Bipolar Depression
Keywords: Depression; MDD; neuroimaging; biomarkers; genomics; proteomic; BP
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression | interventions — Ketamine; Electroconvulsive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Ketamine (Experimental)
  Interventions: Drug: Intravenous Ketamine
- Electroconvulsive Therapy (Active Comparator)
  Interventions: Procedure: Electroconvulsive Therapy

INTERVENTIONS:
Drug: Intravenous Ketamine — Participants will receive 0.5mg/kg IV over 40 minutes, thrice weekly for 3 or 4 weeks. If participant responds, they will receive infusions weekly for one month, once every two weeks for two months, and once every month for three months. Should participant relapse during once monthly dosing, they may return to dosing once every two weeks for the remainder of the study.
  Other Names: Ketalar
  Arms: Intravenous Ketamine
Procedure: Electroconvulsive Therapy — Participants will receive ECT treatment thrice weekly for the 3 or 4 weeks. If participant responds, they will continue to receive ECT, with frequency at the discretion of the treating physician based on best practice guidelines for the remainder of the study.
  Other Names: ECT
  Arms: Electroconvulsive Therapy

SUMMARY:
While there are effective treatments for depression available, some patients do not see results with these options. Often, these patients are referred to electroconvulsive therapy (ECT) which has drawbacks such as adverse side effects, cost, and limited access. Recent research shows that intravenous ketamine may be an alternative option for these patients due to its rapid antidepressant effect sustained with multiple treatments.

This study will recruit 240 participants from the ECT waiting list at the five participating hospitals, and randomize them to either the ketamine or ECT treatment arm. Participants in the ketamine treatment arm will receive 0.5mg/kg ketamine intravenously (IV) over 40 minutes as described in the study schedule. Participants in the ECT treatment arm will receive ECT as described in the study schedule and as decided by their treating physician. Throughout the study, clinical, neuroimaging, molecular, and cognitive assessments will be conducted.

The aim of this study is to show that compared to ECT, ketamine treatment produces faster results, has less side effects, requires less or shorter hospitalizations, and is less expensive. The measures collected throughout the study (clinician scales, self-reports, blood samples, and neuroimaging) may help with predicting if future patients will respond to ECT or ketamine. This could lead to faster, more effective treatment for patient with depression.

DETAILED DESCRIPTION:
Worldwide, depression carries a significant burden. Although there are effective treatments for depression, many patients do not achieve remission, and any significant response usually occurs after a few weeks. The common approach for a rapid intervention in cases of severe depressive symptoms has been electroconvulsive therapy (ECT). There are drawbacks to ECT including a prior medical work-up, general anaesthesia, and the possibility of memory loss. Further, access to ECT is often limited. Comparatively, the most striking breakthrough in the field of mood disorders has been the rapid antidepressant effects of intravenous ketamine. The antidepressant response to ketamine often occurs within a few hours, and peaks within 24. Recent studies have documented that the benefits of ketamine can be sustained with repeated administration.

This longitudinal, multi-centre, randomized, crossover clinical trial is funded in part by the Ontario Brain Institute through a sponsorship with the Canadian Biomarker Integration Network in Depression (CAN-BIND) research program. It will take place across five sites: the Royal Ottawa Mental Health Centre (lead site), Douglas Mental Health University Institute, Providence Care Hospital, Sunnybrook Health Sciences Centre and University Health Network.

A total of 240 participants (accounting for 20% dropout) will be recruited over 30 months from ECT wait lists across the five sites and randomized to either the ketamine or ECT treatment arm. Participants in the ketamine treatment arm will receive 0.5 mg/kg IV over 40 minutes in the recovery room of the ECT clinic as per the study schedule. Participants in the ECT treatment arm will receive ECT as per the study schedule and as decided by their treating physician. Each participant will be enrolled in the study for between six weeks and nine months, or until they leave the study or the study is terminated.

Throughout the study, clinical, neuroimaging, molecular, and cognitive assessments will be conducted. Data will be collected using the Ontario Brain Institute's Centre for Ontario Data Exploration and Research Electronic Data Capture in order to coordinate data from the five sites.

Participants randomized to the either treatment arm will receive thrice weekly treatments for 3 or 4 weeks for a total of 9 or 12 treatments respectively. Following the randomization phase, responders may move to the maintenance phase and non-responders may move to the crossover phase where they will receive the alternate therapy. During the crossover phase, participants will receive thrice weekly treatments for 3 or 4 weeks for a total of 9 or 12 treatments respectively. Following the crossover phase, responders will move to the maintenance phase and non-responders will exit the study. During the maintenance phase, participants who achieved response with ketamine will receive weekly ketamine treatments for one month, treatment once every two weeks for two months, and monthly treatment for three months. Should participants in the ketamine arm relapse during monthly treatment, they may return to treatments once every two weeks. Participants who achieved response in the ECT arm will receive ECT treatment for six months based on decision of the treating physician in order to maintain a clinical response. Both treatment arms will have a follow-up visit during month seven.

The aim of this study is to show that compared to ECT, ketamine treatment produces faster therapeutic action, has less side effects, requires fewer/shorter hospitalizations for patients, and will be less expensive because it does not require an anaesthesiologist and a psychiatrist to administer the various ECT protocols. Through the discovery of biomarkers to predict ECT or ketamine response or non-response, the anticipated effective treatment could be administered as a first line intervention for a subgroup of depressed patients, thereby ensuring a more time-efficient intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent before initiation of any study-related procedures.
2. Eligible subjects who have consented to standard ECT treatment for their mood disorder and are willing to accept randomization to either ECT or IV ketamine group.
3. Men and women aged between 18 and 70 years, inclusive with a body mass index (BMI) < 35. They must have a Montreal Cognitive Assessment (MOCA) score ≥ 24.
4. Patients meeting criteria for Major Depressive Disorder (MDD) or Bipolar Disorder (BP) without psychotic symptoms according to the Diagnostic and Statistical Manual for Mental Disorders (DSM-5) currently in a Major Depressive Episode (MDE) as confirmed by the MINI International Neuropsychiatric Interview (MINI).
5. A Montgomery-Åsberg Depression Rating Scale (MADRS) total score of ≥ 26 at screening and at randomization, with no more than 20% improvement between these two visits.
6. Female subjects of childbearing potential must have a negative urine pregnancy test at enrolment (Visit 1) and be willing to use a reliable method of birth control (i.e., double-barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device, or tubal ligation) during the study.
7. Abstain from consuming grapefruit juice (a potent 3A4 cytochrome inhibitor) on the day of the ketamine infusions as it may slow down the elimination of ketamine.
8. Be able to understand and comply with the requirements of the study, as judged by the investigator(s).

Exclusion Criteria:

1. Depression secondary to stroke, cancer or other severe medical illnesses.
2. Prior or current substance abuse or dependence (except for caffeine or nicotine dependence) and/or recent history (last 12 months) of current alcohol abuse or dependence, as defined in DSM-5 criteria ("a problematic pattern of using alcohol or another substance that results in impairment in daily life or noticeable distress").
3. A positive toxicology screen for drugs that are not prescribed.
4. Unwilling to maintain current antidepressant regimen.
5. Unwilling or unable to hold benzodiazepines from the evening prior to the infusion of ketamine.
6. Unwilling to discontinue any narcotic for a minimum of 5 drug half-lives prior to injections.
7. Pregnant, lactating, or of childbearing potential and not willing to use an approved method of contraception during the study.
8. Evidence of clinically relevant disease, e.g., uncontrolled hypertension, renal or hepatic impairment, significant coronary artery disease (myocardial infarct within a year prior to initial randomization), cerebrovascular disease, history of cerebrovascular accident, viral hepatitis B or C, acquired immunodeficiency syndrome.
9. A clinical finding that is unstable or that, in the opinion of the investigator(s), would be negatively affected by the study medication or that would affect the study medication (e.g., diabetes mellitus, hypertension, unstable angina).
10. Liver function tests AST and ALT three times the upper normal limit at screening.
11. Uncorrected hypothyroidism or hyperthyroidism. Subjects needing a thyroid hormone supplement to treat hypothyroidism must have been on a stable dose of the medication for 30 days prior to enrolment (Visit 1).
12. Clinically significant deviation from the reference range in clinical laboratory test results as judged by the investigator(s). Including:

    * Sodium under 135 or over 145 mmol/L
    * Potassium under 3.5 or over 5.0 mmol/L
    * Chloride under 98 or over 106 mmol/L
    * ALT under 17 or over 63 U/L
    * AST under 18 or over 40 U/L
    * Total bilirubin over 26 mmol/L
    * GGT under 9 or over 48 U/L
    * Fasting glucose under 3.3 or over 5.8 mmol/L
    * BUN under 2.5 or over 8.0 mmol/L
    * Creatinine under 50 or over 90 mmol/L in females, and under 70 or over 120 mmol/L in males
    * TSH under 0.4 or over 5.0 mU/L
    * CBC indicating:
    * Hemoglobin under 123 or over 157 g/L in females, and under 130 or over 170 g/L in males
    * Hematocrit under 0.370 or over 0.460 in females, and under 0.380 or over 0.50 in males
    * RBC under 4.0 or over 5.2x1012/L in females and under 4.4 or over 5.7x1012/L in males
    * MCV under 80 or over 100 fL
    * WBC under 4 or over 10x109/L
    * Neutrophil over 0.7x109/L
    * Lymphocyte under 1.0 or over 4.0x109/L
    * Monocyte under 0.1 or over 1.0x109/L
    * Eosinophil over 0.45x109/L
    * Basophils over 0.10x109/L
    * Platelets under 130 or over 400x109/L
13. ECG results considered clinically significant as determined by the investigator(s), or outside of normal range as per cardiologist analysis.
14. History of seizure disorder, except febrile convulsions.
15. Known history of intolerance or hypersensitivity to ketamine.
16. Any other condition that, in the opinion of the investigator(s), would adversely affect the subject's ability to complete the study or its measure.

Note: active suicidal intent in MDD with the absence of psychotic symptoms is not an exclusion criterion).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | 3-4 weeks
  Change in MADRS (Montgomery-Asberg Depression Rating Scale) scores from baseline.
  * Remission: MADRS ≤ 10
  * Response: >50% reduction in MADRS from baseline and a score <22

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Blier, MD, PhD, Principal Investigator — The Royal's Institute of Mental Health Research
Locations (4):
- Canada (4):
  - Providence Care Hospital, Kingston, Ontario
  - Royal Ottawa Mental Health Centre, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Ontario Shores Centre for Mental Health Sciences, Whitby, Ontario

IPD SHARING:
Plan to Share IPD: Yes
This study is funded by the Ontario Brain Institute (OBI). Data collected from this study is entered into a research database called "Brain-CODE", deployed at a High Performance Computer Virtual Lab (HPCVL). The HPCVL supports the regulatory-compliant (e.g. 21 CRF Part 11, HIPPA, PIPEDA) processes for securing privacy of healthcare data.

REFERENCES:
- [Derived] Phillips JL, Jaworska N, Kamler E, Bhat V, Blier J, Foster JA, Hassel S, Ho K, McMurray L, Milev R, Moazamigoudarzi Z, Placenza FM, Richard-Devantoy S, Rotzinger S, Turecki G, Vazquez GH, Kennedy SH, Blier P; CAN-BIND Investigator Team. A randomized, crossover comparison of ketamine and electroconvulsive therapy for treatment of major depressive episodes: a Canadian biomarker integration network in depression (CAN-BIND) study protocol. BMC Psychiatry. 2020 Jun 2;20(1):268. doi: 10.1186/s12888-020-02672-3. PMID 32487236